CLINICAL TRIAL: NCT04801433
Title: A Multicenter, Randomized, Single-blind, Parallel-controlled Clinical Study to Evaluate the Efficacy and Safety of Boroda Supramolecular Active Zinc in the Treatment of Scalp Psoriasis
Brief Title: Evaluate the Efficacy and Safety of Boroda Supramolecular Active Zinc in the Treatment of Scalp Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Gang Wang, MD, chief of dermatology, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XijingH-PF-Pso-2018/2019
Record Dates: First submitted 2021-03-09; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Scalp Psoriasis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Boleda Supramolecular Active Zinc (Experimental): Boleda Supramolecular Active Zinc (Shanghai Ruizhi Pharmaceutical Technology Co., Ltd.): 30ml/bottle. Once a day for 4 weeks, apply topically to the scalp psoriasis area, gently massage for 15 minutes then rinse off with warm water.
  Interventions: Other: Boleda Supramolecular Active Zinc Conditioner
- Capotetriol scalp solution (Active Comparator): 30ml/bottle. Two times a day for 4 weeks, topically applied to scalp psoriasis.
  Interventions: Drug: Capotetriol scalp solution
- Supramolecular Hydrogel (Placebo Comparator): 30ml/bottle. Once a day for 4 weeks, apply topically to the scalp psoriasis area, gently massage for 15 minutes then rinse off with warm water.
  Interventions: Other: Supramolecular Hydrogel

INTERVENTIONS:
Other: Boleda Supramolecular Active Zinc Conditioner — Boleda Supramolecular Active Zinc Conditioner (Shanghai Ruizhi Pharmaceutical Technology Co., Ltd.): 30ml/bottle. Once a day for 4 weeks, apply topically to the scalp psoriasis area, gently massage for 15 minutes then rinse off with warm water.
  Arms: Boleda Supramolecular Active Zinc
Drug: Capotetriol scalp solution — Capotetriol scalp solution: 30ml/bottle. Two times a day for 4 weeks, topically applied to scalp psoriasis.
  Arms: Capotetriol scalp solution
Other: Supramolecular Hydrogel — Supramolecular Hydrogel (Shanghai Ruizhi Pharmaceutical Technology Co., Ltd.): 30ml/bottle. Once a day for 4 weeks, apply topically to the scalp psoriasis area, gently massage for 15 minutes then rinse off with warm water.
  Arms: Supramolecular Hydrogel

SUMMARY:
A multicenter, randomized, single-blind, parallel-controlled clinical study to evaluate the efficacy and safety of boroda supramolecular active zinc in the treatment of scalp psoriasis.

Main objective:：Compare the efficacy of boroda supramolecular active zinc and capotetriol liniment in the treatment of scalp psoriasis Secondary objective: To observe the safety of boroda supramolecular active zinc in the treatment of subjects with scalp psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-65，regardless of gender；
2. Clinically diagnosed as scalp psoriasis and severity of the disease：

   * According to the researchers evaluation of clinical signs, each of the three clinical signs of scalp psoriasis, erythema, infiltration and scales, needs to be < 3 points, and at least one sign score is ≥ 1.
   * <25% of the total scalp area (the fully expanded flat palm (including the surface of five fingers) is equivalent to approximately 25% of the scalp area).
   * The judgment of mild to moderate outcome need to be in accordance with the overall evaluation criteria;
3. At the time of admission, the skin lesions of the body and limbs of the subjects need to have clinical signs of psoriasis vulgaris (the maximum surface of the affected area is ≤10%) or had been diagnosed as psoriasis vulgaris on the body and limbs at the early stage.
4. Subjects must sign a informed consent of notification in prior to the study;

Exclusion Criteria:

1. Subjects are diagnosed with active guttate psoriasis, pustular psoriasis, arthropathy psoriasis and erythroderma psoriasis at present.
2. The subjects scalp associated with other diseases that may affect the judgment of curative effect: such as, viral infection, fungal infection, bacterial infection, parasitic infection, skin manifestations associated with syphilis or tuberculosis, rosacea, acne, post-acne inflammation, skin atrophy, atrophic stria, increased skin venous vulnerability, ichthyosis, ulcer or wound that skin manifestations related to injury;
3. Any infectious skin disease that confuses the evaluation of the efficacy of scalp psoriasis
4. The subjects that had received systemic biotherapy (listed or not listed) in the past three months of randomized enrollment that may have potential effects on scalp psoriasis, such as alefaxer, legalizumab, etanercept, infliximab, etc.
5. The subjects who had received non-biological systemic therapies that may have an impact on scalp psoriasis, such as corticosteroids, vitamin D-type drugs, Tretinoin, immunosuppressive agents, etc. in 4 weeks before the 2nd screening visit or during the study period.
6. Randomly enrolled (1st visit) subjects who have received PUVA treatment 4 weeks before or during the study period;
7. Randomly enrolled (1st visit) subjects that had received ultraviolet therapy 2 weeks before or during the study period;
8. The subjects that had received the following treatments 2 weeks before the 2nd screening or during the study period:

   1. Strong or extremely effective steroid hormone external preparations for psoriasis on the body and limbs (WHO Class III-IV);
   2. External immunomodulators (such as tacrolimus ointment, etc.)
   3. External use of vitamin D analogues (e.g. captopril preparation, tacalcitol and calcitriol);
   4. External treatment of various types of scalp psoriasis (except for shampoos or softeners that are not steroid drugs);
   5. Other treatments for psoriasis: such as traditional Chinese medicine or Chinese patent medicine, hot springs, etc.
9. During the study period, it is planned to start or change the use of concomitant drugs that may affect scalp psoriasis, such as beta-blockers, antimalarials, lithium preparations, etc.
10. Subjects who are known or suspected to be allergic to the drug components in the study;
11. Pregnant or fertile female intend to be pregnant or lactating during the study period;
12. In the 2nd screening visit, the serum or urine pregnancy test of fertile women is positive.
13. The subjects who participated in other clinical trials within 4 weeks of randomization;
14. The subjects with known or suspected poor compliance who could not complete the tests, such as alcoholism, drug dependence or mental illness, or the subjects who are not suitable to participate in this clinical research that determined by the researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Success rate at the end of treatment (4th week) in each group (percentage of patients with overall score of < 1) | Change of success rate from baseline at 4 weeks
  The overall criteria for assessing the severity of disease for researchers are a static skin scoring system consisting of six levels (score of 0-5) of change from "disappearance" to "very serious" diseases.
  The main endpoint of the overall assessment criteria for disease severity according to the researchers will be "disease control", defined as "disappearance (score of 0) " or "extreme mild (score of 1) " disease grade at the end of treatment.
  At the end of treatment, the proportion of the subjects who are evaluated as disease under control (signs disappeared and extremely mild) by "the overall assessment of the severity of disease by researchers" base on observation. Comparing the disease control rates among the groups can reflect the differentiation treatment efficacy.
The clinical signs of psoriasis (erythema, infiltration, and scaly) (The Total sign score (TSS)) | Change of sclinical signs of psoriasis from baseline at 4 weeks
  Scoring each symptom once on the basis of the five-point system given below can assess the average severity of all scalp lesions.
  0 = no sign
  1. = Mild
  2. = Medium
  3. = Severity
  4. = Extremely severe
  At the end of treatment, researchers need to evaluate scalp psoriasis in all subjects from three aspects: erythema, infiltration and scales. The percentage of remission per clinical sign (erythema, infiltration, scales) in each group (percentage of patients with clinical score = 0).

SECONDARY OUTCOMES:
Evaluation criteria of pruritus symptoms in the subjects | Change of spruritus symptoms from baseline at 4 weeks
  At the end of treatment, the subject are assessed for the severity of the disease according to the four-level system presented below. Researchers should explain the grading criteria to patients, and the subjects should judge the grading and tick it.
  1. Asymptomatic: no itching;
  2. Mild: mild itching, no irritation;
  3. Moderate: markedly itchy, somewhat irritable, but no insomnia;
  4. Severe: Strong itching causes significant irritability, affects sleep, and scratches are visible.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Derpartment of Xijing Hospital, Xi'an, Shaanxi, China